CLINICAL TRIAL: NCT04498403
Title: A PHASE 3, MULTICENTER, OPEN-LABEL STUDY OF THE LONG-TERM SAFETY OF CRISABOROLE OINTMENT, 2% IN JAPANESE PEDIATRIC AND ADULT PARTICIPANTS WITH MILD TO MODERATE ATOPIC DERMATITIS
Brief Title: A Study of the Long-Term Safety of Crisaborole Ointment, 2% in Japanese Pediatric and Adult Participants With Mild to Moderate Atopic Dermatitis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Terminated (This decision was made for business reasons only and is not related to any safety concerns regarding crisaborole.)
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C3291027
Record Dates: First submitted 2020-07-31; First posted 2020-08-04 (Actual); Results first posted 2021-08-12 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-07

CONDITIONS: Atopic Dermatitis
Keywords: Eczema; Crisaborole
MeSH Terms: conditions — Dermatitis, Atopic; Eczema

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Crisaborole 2% (Experimental): Crisaborole 2% ointment applied twice daily (BID)
  Interventions: Drug: Crisaborole 2%

INTERVENTIONS:
Drug: Crisaborole 2% — Crisaborole 2% ointment

SUMMARY:
This study is a Phase 3, multicenter, open-label, long-term safety extension study of Studies C3291032 and C3291031 in Japanese pediatric and adult participants with mild to moderate Atopic Dermatitis (AD).

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants;
* Who were patients with mild to moderate AD aged 2 years old or older and met eligibility criteria for study C3291032 at the time when entering Study C3291032, and completed treatment period in Study C3291032 without safety issues. Or
* Who were patients with mild to moderate AD aged 1 months to <24 months and met eligibility criteria for Study C3291031 at the time when entering Study C3291031, and completed treatment period in Study C3291031 without safety issues

Exclusion Criteria:

* Has other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.

Min Age: 7 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2020-12-18 (Actual); Study Completion 2020-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (11):
- Japan (11):
  - Shirao Clinic of Pediatrics and Pediatric Allergy, Hiroshima, Hiroshima
  - Chitose dermatology and plastic surgery clinic, Chitose Shi, Hokkaido
  - Takagi Dermatological Clinic, Obihiro, Hokkaido
  - Yoshimura Child Clinic, Akashi, Hyōgo
  - Iryouhoujinshadan Yamayurikai Tsujino. Kodomo Clinic, Kobe, Hyōgo
  - Noguchi Dermatology Clinic, Kamimashiki-gun, Kumamoto
  - Yoshioka Dermatology Clinic, Neyagawa, Osaka
  - Mildix Skin Clinic, Adachi-ku, Tokyo
  - Yoga Allergy Clinic, Setagaya-ku, Tokyo
  - Sugamo Kobayashi Derma Clinic, Toshima-Ku, Tokyo
  - Hoshikuma Dermatology・Allergy Clinic, Fukuoka

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3291027

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: Crisaborole 2%, Age Group: Less Than (<) 18 Years: Participants aged < 18 years with mild to moderate atopic dermatitis (AD) received crisaborole ointment, 2 percent (%) on treatable AD lesions, twice daily. Treatable AD lesions were identified at Baseline (Day 1) by investigator. Participants were followed up to at least 28 days after last dose of study drug.
- Cohort 2: Crisaborole 2%, Age Group: Greater Than or Equal to (>=) 18 Years: Participants aged >= 18 years with mild to moderate atopic dermatitis (AD) received crisaborole ointment, 2 percent (%) on treatable AD lesions, twice daily. Treatable AD lesions were identified at Baseline (Day 1) by investigator. Participants were followed up to at least 28 days after last dose of study drug.
Period: Overall Study
Arm/Group | Cohort 1: Crisaborole 2%, Age Group: Less Than (<) 18 Years | Cohort 2: Crisaborole 2%, Age Group: Greater Than or Equal to (>=) 18 Years
Started | 30 | 10
Completed Follow up | 30 | 10
Completed | 0 | 0
Not Completed | 30 | 10
Not completed — Adverse Event | 1 | 0
Not completed — Study Terminated By Sponsor | 29 | 10

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who took at least 1 dose of study drug. Participants who entered the first Off-Treatment cycle were included.
Groups:
- Cohort 1: Crisaborole 2%, Age Group: Less Than (<) 18 Years: Participants aged < 18 years with mild to moderate AD received crisaborole ointment, 2 % on treatable AD lesions, twice daily. Treatable AD lesions were identified at Baseline (Day 1) by investigator. Participants were followed up to at least 28 days after last dose of study drug.
- Cohort 2: Crisaborole 2%, Age Group: Greater Than or Equal to (>=) 18 Years: Participants aged >= 18 years with mild to moderate AD received crisaborole ointment, 2 % on treatable AD lesions, twice daily. Treatable AD lesions were identified at Baseline (Day 1) by investigator. Participants were followed up to at least 28 days after last dose of study drug.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Crisaborole 2%, Age Group: Less Than (<) 18 Years | Cohort 2: Crisaborole 2%, Age Group: Greater Than or Equal to (>=) 18 Years | Total
Number analyzed (Participants) | 30 | 10 | 40
Age, Continuous [Mean (Standard Deviation); unit: Years] | 9.3 (3.99) | 31.8 (7.97) | 15.0 (11.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 4 | 19
  Male | 15 | 6 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 30 | 10 | 40
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 30 | 10 | 40
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An adverse events (AE) is any untoward medical occurrence in clinical investigation participant administered a product or medical device; event need not necessarily to had a causal relationship with treatment or usage. SAEs: an AE resulting in any of following outcomes/deemed significant for any other reason: death; initial/prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. TEAEs are events between first dose of study drug and up to 28 days after last dose of study drug, that were absent before treatment or that worsened relative to pretreatment state. AEs included both serious and non-serious adverse events.
Time Frame: Baseline up to 28 days after last dose of study drug (maximum up to 12 weeks)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Crisaborole 2%, Age Group: Less Than (<) 18 Years | Cohort 2: Crisaborole 2%, Age Group: Greater Than or Equal to (>=) 18 Years
Number analyzed (Participants) | 30 | 10
Participants
  TEAEs | 11 | 3
  SAEs | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to 28 days after last dose of study drug (maximum up to 12 weeks)
Arm/Group | Cohort 1: Crisaborole 2%, Age Group: Less Than (<) 18 Years | Cohort 2: Crisaborole 2%, Age Group: Greater Than or Equal to (>=) 18 Years
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/10
Other Adverse Events (participants affected / at risk) | 11/30 | 3/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Crisaborole 2%, Age Group: Less Than (<) 18 Years (N=30) | Cohort 2: Crisaborole 2%, Age Group: Greater Than or Equal to (>=) 18 Years (N=10)
Application site pain (General disorders) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Molluscum contagiosum (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 3 | 0
Otitis media acute (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 2 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Participants were planned to be followed up to Week 56, however due to early termination of the study, participants were followed up to only Week 12.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2020-05-20): https://cdn.clinicaltrials.gov/large-docs/03/NCT04498403/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-07): https://cdn.clinicaltrials.gov/large-docs/03/NCT04498403/SAP_001.pdf